CLINICAL TRIAL: NCT07076264
Title: Water Competency Intervention for Children on the Autism Spectrum: The AquOTic Hybrid Effectiveness Implementation Trial
Brief Title: Water Competency Intervention in Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jewel Crasta, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20250101; E06288.1a (Other Grant/Funding Number: Congressionally Directed Medical Research Program)
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorders
Keywords: Swim Safety; Water Competency; Occupational Therapy; AquOTic; Drowning Prevention
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study employs a hybrid Type I efficacy-implementation design, aiming to evaluate both the effectiveness of the AquOTic intervention and to advance the science of implementation. While hybrid Type I trials traditionally emphasize clinical effectiveness, this study extends beyond identifying implementation barriers and facilitators by preliminarily assessing proposed implementation mechanisms. Specifically, it will examine therapeutic alliance and attitudes toward the AquOTic intervention as hypothesized factors associated with high intervention fidelity. The trial will utilize a single-blinded, randomized controlled trial (RCT) design, with participants randomly assigned to one of three study arms: (1) AquOTic with professional student interventionists, (2) AquOTic with community interventionists, or (3) a control group receiving no AquOTic intervention, while outcomes assessors will remain blinded to group assignment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AquOTic with Professional Student Interventionist (Experimental): Participants in this arm will participate in the 10-week AquOTic intervention with their one to one interventionists being professional students (OT/PT students currently enrolled at OSU).
  Interventions: Other: AquOTic
- AquOTic with Community Interventionists (Experimental): Participants in this arm will participate in the 10-week AquOTic intervention with their one to one interventionists being community interventionists (high school or undergraduate students in the community).
  Interventions: Other: AquOTic
- Control Group (No Intervention): Participants will NOT receive AquOTic intervention and will engage in usual and customary water exposure.

INTERVENTIONS:
Other: AquOTic — AquOTic is an evidence-based, occupational therapy-led intervention designed to enhance water competency and swim safety skills in children on the autism spectrum. The 10-week program consists of weekly 60-minute group sessions, each including six children paired in a 1:1 ratio with an interventionist. Sessions follow a structured routine involving six rotating stations, targeting various swim and safety skills, with the flexibility for individualized support by the interventionist.
  Arms: AquOTic with Community Interventionists; AquOTic with Professional Student Interventionist

SUMMARY:
AquOTic is an evidence-based, occupational therapy-led intervention designed to enhance water competency and swim safety skills in children on the autism spectrum. The 10-week program consists of weekly 60-minute group sessions, each including six children paired in a 1:1 ratio with an interventionist. Sessions follow a structured routine involving six rotating stations, targeting various swim and safety skills, with the flexibility for individualized support by the interventionist.

Overall, this study has 3 major aims. The first aim evaluates the effectiveness of the AquOTic intervention in improving water competency and swim skills, while comparing outcomes between two implementation models: professional student interventionists (occupational and physical therapy students) and trained community-based interventionists. A total of 108 autistic children will be enrolled and randomly assigned to one of three groups: (1) AquOTic with professional student interventionists, (2) AquOTic with community interventionists, or (3) a control group receiving no AquOTic intervention. The second aim explores the mediators and moderators of the intervention outcomes to assess fidelity and efficacy. The third aim identifies the cost and resources associated with AquOTic. A cost analysis will be conducted to evaluate the resources required for implementation and to inform the development of a scalable, cost-effective drowning prevention strategy for autistic populations.

ELIGIBILITY:
Children Participants (n=108)

Inclusion Criteria

* Educational or medical diagnosis of autism
* Age between 5 - 9 years
* Having vision and hearing within normal limits with or without corrective modifications

Exclusion Criteria

* Children who demonstrate swim proficiency, as defined by the ability to tread water for 1 minute or move the body through the water without flotation
* Open wounds or infectious skin diseases
* Allergy to chlorine
* Severe co-occurring motor impairments or neurological conditions such as uncontrolled seizures, Rett's or Angelman's syndrome
* The family is unable to commit to the sessions or evaluations

Interventionists (n=64)

Inclusion Criteria

* Aged 18 or over
* Demonstrate swim proficiency, as defined by the ability to tread water for 1 minute and move the body through the water without flotation for 25 yards

Exclusion Criteria

* Open wounds or infectious diseases
* Failed background check
* Unable to commit to Basic Swim Instructor and AquOTic training (~40 hours) and 10 AquOTic sessions (20 hours)

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Water Orientation Test-Alyn (WOTA) 2 | At baseline, immediately post-AquOTic, 6 months after termination of AquOTic, and 12 months after termination of AquOTic
  The WOTA2 measures a child's mental adaptation, adjustment to the pool, postural balance, and the ability to move and change position in the water, based on the Halliwick concept. WOTA2 assesses 27 swim skills scored on a 0-3 scale with a minimal detectable change score of 11.5. Higher scores indicate better skills. WOTA2 has high test-retest reliability (ICC=.97) and is validated for children with autism-like characteristics.

SECONDARY OUTCOMES:
Water Orientation Test-Alyn (WOTA) 1 | At baseline, immediately post-AquOTic, 6 months after termination of AquOTic, and 12 months after termination of AquOTic
  WOTA1 measures a child's mental adaptation, adjustment to the pool, postural balance, and the ability to move and change position in the water, based on the Halliwick concept. WOTA1 assesses 13 swim skills on a 1-4 scale with a minimal detectable change score of 4.5.
Water Competency Checklist (WCC) | At baseline, immediately post-AquOTic, 6 months after termination of AquOTic, and 12 months after termination of AquOTic
  WCC was developed by the AquOTic team and incorporates additional skills not on the WOTA that are considered necessary for water competence. These include jumping in and resurfacing, treading water, and turning around in the water. This checklist is a compilation of items from other swim checklists such as those used by the American Red Cross and clinical trials of swim interventions in autism
Canadian Occupational Performance Measure (COPM) | At baseline, immediately post-AquOTic, 6 months after termination of AquOTic, and 12 months after termination of AquOTic
  COPM is an individualized standardized outcome measure sensitive to change in performance over time. The COPM has been adapted for use in pediatric clinical trials for caregivers of children with disabilities. This measure will be administered by an occupational therapist via a semi-structured interview in which caregivers will identify 3-5 functional goals related to swim performance and water safety. Caregivers will rate how well their child performed each goal (COPM - Performance), and how satisfied they are with their child's performance (COPM - Satisfaction). The same caregiver will be interviewed at pre- and post-test assessments for the AquOTic program. A change of 2 or more points in each scale of the COPM is considered a minimum clinically important difference (MCID). The adapted COPM has high internal consistency (.86 - .88) with content and construct validity.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data on outcome measures with the NIH National Database of Autism Research (NDAR). A README file and data dictionary will be generated and deposited into the NDA repository along with all shared datasets to facilitate the interpretation and reuse of the data. The README file will include the study protocol and data dictionary. All data will be de-identified prior to receipt by the repository, but the information needed to generate a global unique identifier (GUID) will be collected for each participant. During study enrollment, we will collect name, date of birth, gender, and town/municipality of birth for all participants to facilitate the creation of a GUID for each participant. Information about NDA data sharing will be included in the consent documentation for the study to allow participants to choose whether they wish to consent to data sharing through NDA.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified data will be made available after the completion of the study.

REFERENCES:
- [Result] Kemp E, Nikahd M, Howard M, Darragh A, Crasta JE. Improving water competency among children on the autism spectrum: the AquOTic randomized controlled trial. Front Pediatr. 2024 Oct 7;12:1473328. doi: 10.3389/fped.2024.1473328. eCollection 2024. PMID 39435387